CLINICAL TRIAL: NCT06265337
Title: Does Co-administration of Lactate to an Oral Glucose Tolerance Test Lower the Glucose Response?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Natasa Brkovic Zubanovic, Principal investigator, M.D, Phd-student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LAMETA-OGTT
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-02

CONDITIONS: PreDiabetes; Metabolic Syndrome; Insulin Resistance
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome; Insulin Resistance | interventions — Lactic Acid

STUDY DESIGN:
Intervention Model Description: In a randomized, double-blinded, placebo-controlled crossover trial, we will investigate the effect of addition of 25 g lactate vs. placebo to an OGTT on two trial days separated by a minimum of fourteen days and a maximum of one month. We will include 12 individuals with pre-diabetes [9], having HbA1c 39-47 mmol/L and being above 40 years of age.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAC (Experimental)
  Interventions: Dietary Supplement: Lactate; Other: Placebo
- CTR (Placebo Comparator)
  Interventions: Dietary Supplement: Lactate; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactate — Lactate in an OGTT (300 mL lactate drink = 25 g D/L-lactate bound to Na) =LAC with a stable isotope glucose tracer (D2-glucose) added to measure glucose.
Other: Placebo — Placebo in an OGTT (300 mL salt water, NaCl) =CTR with a stable isotope glucose tracer (D2-glucose) added to measure glucose.

SUMMARY:
To investigate whether co-administration of lactate with a glucose load affects postprandial glucose levels/handling, gastrointestinal hormones, gastric emptying, and appetite sensations in individuals with pre-diabetes when compared to placebo.

Hypothesis:

Oral lactate administration improves/lowers glucose excursions following an oral glucose tolerance test (OGTT) by stimulating insulin secretion and delaying glucose absorption.

DETAILED DESCRIPTION:
The participants will be instructed to avoid hard-to-moderate physical activity for 48 hours before each of the two trial days. They will be instructed to eat the same diet 72 hours before the two trial days at the screening visit and to register it in MyFood24 which is an electronic foodlog.

Trial days:

The two trial days will be completely alike, besides the interventions consisting of either:

1. Placebo in an OGTT (300 mL salt water, NaCl) =CTR, or
2. Lactate in an OGTT (300 mL lactate drink = 25 g D/L-lactate bound to Na) =LAC with a stable isotope glucose tracer (D2-glucose) added to each of the interventions to measure glucose uptake. 1500 mg of paracetamol will be added to measure ventricular emptying rate using the acetaminophen test.

An H3-glucose tracer will be continuously infused to measure glucose turnover. Glucose tolerance and absorption together with hepatic glucose production and insulin secretion will be quantified using the oral minimal model.

After this, the participant can lie in their bed. Blood samples will be collected continuously during the day. Appetite sensations will be measured by a visual analogue scale (VAS). After 4 hours the trial day is finished, and the participants can go home.

They will be instructed to collect two fecal samples after each of the trial days, which will be analysed for fecal microbiota composition (16S rRNA gene sequencing and quantitative PCR) and fecal fermentation metabolite profiles by our collaborator Clarissa Schwab.

Analyses Blood sample analyses will be made for the concentration of lactate, insulin, GLP-1, GIP, ghrelin, LEAP-2, glucagon, c-peptide, blood glucose, triglycerides, cholesterol, and other relevant metabolites and hormones. Supplementary ventricular emptying rate will be compared between CTR and LAC. [3H ]-glucose-tracer will be infused for six hours (bolus 12 mCi, infusion 0,12 mCi/min) to determine glucose metabolism.

Statistics and power calculation We will use simple paired t-tests and two-way repeated measure ANOVA analyses for comparing the two groups.

Based on a previous study we will need 12 individuals to detect a difference of 15% in integrated glucose concentrations and 40% in disposition index after the OGTT (α=0.05, β=0.80). This is similar to the effect size observed in studies investigating the treatment with a dipeptidyl peptidase-4 inhibitor (a weak insulin secretagogue).

ELIGIBILITY:
Inclusion Criteria:

* >40 years

  * Written and oral consent
  * HbA1c 39-47 mmol/L

Exclusion Criteria:

* Medicine with an impact on blood glucose and glucose metabolism
* Newly started medicine (<3 months prior to the inclusion time)
* Medicine changes (<3 months prior to the inclusion time and planned changes during the trial)
* Affected screening blood sample as evaluated by PI
* Hba1c > 47
* Allergy to paracetamol
* Doesn't speak or understand Danish.
* Special diets

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Difference in integrated glucose concentrations between CTR and LAC following an OGTT | 0-240 minutes after the OGTT

SECONDARY OUTCOMES:
Difference in glucose absorption | 0-240 minutes after the OGTT
  Oral minimal model
Difference in insulin sensitivity | 0-240 minutes after the OGTT
  Oral minimal model
Difference in insulin secretion | 0-240 minutes
  Oral minimal model
Difference in free fatty acids concentration | 0-240 minutes after the OGTT
Difference in ventricular emptying rate | 0-240 minutes after the OGTT
  Acetaminophen test
Difference in subjective appetite sensation | 0-240 minutes after the intervention
  VAS score
Difference in integrated GLP-1 concentrations | 0-240 minutes after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Esben Søndergaard, Principal Investigator — Aarhus University, Steno Diabetes Center Aarhus
Locations (1):
- Steno Diabetes Centre, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided